CLINICAL TRIAL: NCT07002398
Title: A Single Arm, Ph1/2, Open-label, Multicenter Trial With Dose-exploration Via Subretinal Injection to Evaluate the Safety and Preliminary Efficacy of VG801 for Treatment of ABCA4 Mutation-associated Recessive Hereditary Retinal Dystrophy (Stargardt Disease)
Brief Title: Safety and Preliminary Efficacy of VG801 in Patients With ABCA4 Mutation-associated Retinal Dystrophy (Stargardt Disease)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VeonGen Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VG801-2022A
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-01

CONDITIONS: Retinal Dystrophy Due to Biallelic ABCA4 Mutations; Stargardt Disease 1
Keywords: ABCA4 mutation; Gene therapy; Eye disease; Stargardt disease; Retinal disease; Retinal degeneration; VG801
MeSH Terms: conditions — Stargardt Disease; Eye Diseases; Retinal Diseases; Retinal Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- VG801 (Experimental): Participants will receive a single dose of subretinal injection of VG801at Day 0.
  Interventions: Drug: VG801

INTERVENTIONS:
Drug: VG801 — Administered as specified in the single treatment arm. Study Cohort: Low dose, medium dose and high dose cohort

SUMMARY:
This is a single-arm, open-label, non-randomized, single dose-escalation, first-in-human (FIH) clinical trial to evaluate the safety and preliminary efficacy of VG801 for treatment of patients with retinal dystrophy (Stargardt disease) due to biallelic ABCA4 mutations.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for study entry, subjects must satisfy all the following criteria:

1. Written informed consent.
2. Subjects aged ≥ 6 years.
3. Clinical diagnosis of a macular lesion phenotypically consistent with a recessive hereditary macular dystrophy (Stargardt disease).
4. Confirmed molecular diagnosis of ABCA4 mutations (homozygotes or compound heterozygotes).
5. Poor vision in the study eye.

Exclusion Criteria:

Subjects will be excluded from the study if one or more of the following statements are applicable to either eye:

1. Pre-existing eye conditions such as uveitis, glaucoma, or diabetic retinopathy or implantation of a medical device in the vitreous cavity or subretinal space.
2. Systemic diseases that would preclude the planned surgery or interfere with the interpretation of study results.
3. History of intraocular surgery within the previous 6 months.
4. Previous participation in a gene therapy trial.
5. Participation in a clinical trial (investigational drug or medical device) within the previous 6 months.
6. Any other eye disease that may affect the outcome of the study (e.g., ocular opacities, advanced cataracts, amblyopia, etc.).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline to Month 12
  Abnormal examination results will be recorded.

SECONDARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | Screening to Month 12
  Abnormal examination results will be recorded.
Optical coherence tomography (OCT) | Baseline to Month 12
  Abnormal examination results will be recorded.
Fundus autofluorescence | Baseline to Month 12
  Abnormal examination results will be recorded.
Microperimetry | Baseline to Month 12
  Abnormal examination results will be recorded.
Novel Virtual Reality Visual Test (Exploratory) | Baseline to Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Sun, MD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided